CLINICAL TRIAL: NCT03971240
Title: Traumatic Acute Subdural Haematoma: Management and Outcome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Ahmed Ibrahim Alghriany, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: acute subdural hematoma
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Traumatic Brain Hemorrhage
MeSH Terms: conditions — Brain Hemorrhage, Traumatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- outcome of surgically evacuated traumatic ASDH (Experimental): we will operate patients with traumatic acute subdural hematoma with some criteria and evaluate the outcome of surgery
  Interventions: Procedure: evacuation of traumatic acute subdural hematoma

INTERVENTIONS:
Procedure: evacuation of traumatic acute subdural hematoma — craniotomy will be done with evacuation of the hematoma

SUMMARY:
Traumatic acute subdural haematomas (ASDHs) are common pathological entity in neurosurgical practice . The frequency of (ASDHs) has been proposed as approximately 10-20% of patients admitted with traumatic brain injury(TBI) .Approximately two -thirds of patient with TBI undergoing emergency cranial surgery have an acute subdural haematoma evacuated . Two common causes of traumatic ASDH: accumulation of blood around parenchymal laceration , usually frontal and temporal lobes and there is usually severe underlying brain injury .The second cause is surface or bridging vessel torn from cerebral acceleration - deceleration during violent head motion .

DETAILED DESCRIPTION:
Traumatic acute subdural haematomas (ASDHs) are common pathological entity in neurosurgical practice . The frequency of (ASDHs) has been proposed as approximately 10-20% of patients admitted with traumatic brain injury(TBI) .Approximately two -thirds of patient with TBI undergoing emergency cranial surgery have an acute subdural haematoma evacuated . Two common causes of traumatic ASDH: accumulation of blood around parenchymal laceration , usually frontal and temporal lobes and there is usually severe underlying brain injury .The second cause is surface or bridging vessel torn from cerebral acceleration - deceleration during violent head motion . These haematomas have been historically associated with high mortality rate (between 40-60%)(1).This high mortality rate has been attributed to the characteristic of haematoma itself , due to the primary insults to the brain like brain parenchymal injury , and to the secondary insults like hypoxia and hypotension in severe head injury patients .

Theoretically ,intracranial hypertension due to ASDH may lead to transtentorial cerebral herniation and secondary ischemic injury of the brain.CT scan is main and most informative investigatory aid in diagnosis of traumatic ASDH. The criteria used to select patients for non - operative management are clinical stability or improvement during the time from injury to evaluation at hospital , haematoma thickness less than 10 mm and mid line shift less than 5 mm in the initial CT. Surgery is indicated if on CT 1- ASDH with thickness > 10mm. or 2- Mid line shift >5mm.on CT 3- ASDH with thickness <10 mm and midline shift <5mm on CT should undergo surgical evaluation if (a) GCS drop by >_ 2 point from injury to admission .(b) and or pupils are asymmetric or fixed and dilated (7). Time of surgery for ASDH is matter of controversy. As general principle ,when surgery for ASDH is indicated it should be done as soon as possible . Regarding evacuation of acute subdural haematoma, procedures vary from single burrhole evacuation to craniotomies and decompressive procedures .Some advocated ASDH evacuations by decompressive craniectomy with dural - slits .

ELIGIBILITY:
Inclusion Criteria:

* patients with traumatic ASDH with thickness greater than 10 mm on CTscan
* patients with traumatic ASDH associated with mid -line shift more than 5 mm on CT scan.

Exclusion Criteria:

* patients with blood diseases or defective coagulation.
* CT demonstrates associated other intracranial hematomas e.g. epidural , intracerebral or subarachenoid haemorrhage.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2020-08-31 (Estimated); Study Completion 2021-01-31 (Estimated)

PRIMARY OUTCOMES:
clinical outcome | within 6 weeks post operative
  evaluation of the clinical outcome by recording the the patients' outcome by modified rankin scale: G"0'' No disability at all. (+1) No significant disability despite symptoms, able to carry out all usual duties and activities.
  (+2) Slight disability ,unable to carry out all previous activities, but able to look after own affairs without assistance.
  (+3) Moderate disability, requiring some help, but able to walk without assistance.
  (+4) Moderately severe disability, unable to walk and attend to bodily needs without assistance.
  (+5) Severe disability, bedridden, incontinent and requiring constant nursing care attention.
  (+6) Dead
radiological outcome | one day post operative and within 6 weeks post operative
  radiological outcome assessment by CT brain scan by measuring the midline shift in millimeters ( mild midline shift if < 5mm , moderate if = 5 mm. and severe midline shift if > 5mm. )

CONTACTS AND LOCATIONS:
Overall Officials: mohamed alghriany, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No